CLINICAL TRIAL: NCT01197703
Title: European Cardio CT Registry
Brief Title: European Cardio Computer Tomography Registry
Status: Completed | Type: Observational
Sponsor: Stiftung Institut fuer Herzinfarktforschung (Other)
Responsible Party: Sponsor
Other Study IDs: Euro CT
Record Dates: First submitted 2010-09-07; First posted 2010-09-09 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-03

CONDITIONS: Consecutive Patients Undergoing Computed Tomography of the Heart for Clinical Indications
Keywords: Clinical Practice Cardiac CT; Clinical Implications Coronary CT Angiography; Radiation Exposure of Coronary CT Angiography; Registry

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The European Cardiac CT Registry has the unique potential to provide important data that will help to clarify the clinical role of cardiac computed tomography (CT), to create guidelines and recommendations for its use, and to identify the most important areas that require specific further research.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion of all consecutive patients with accomplished or attempted CT imaging of the heart (whether imaging of the coronary arteries or other structures of the heart)
* Informed consent to be entered in the registry.
* Inclusion of all consecutive patients with accomplished or attempted coronary CT angiography.
* Inclusion of all patients who undergo coronary CT angiography for clinical indications, with separate analysis of patients with suspected coronary artery disease and previously known coronary artery disease.

Exclusion Criteria:

- Besides the absence of informed consent, and cardiac CT studies performed as part of a research protocol, no exclusion criteria exist.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients that are studies by computed tomography of the heart for clinical indications
Sampling Method: Non-Probability Sample
Enrollment: 7115 (Actual)
Dates: Start 2010-06 (Actual); Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
collect data | June 2009-
  The general aim of the Registry is to collect data from a large number of patients regarding the indications, general use, safety, and therapeutic implications of cardiac CT in European clinical practice.

SECONDARY OUTCOMES:
effect of coronary CT angiography | June 2009-
  A first specific aim of the Registry is the analysis of the effect of coronary CT angiography on downstream resource utilization, revascularization procedures, and prognosis in patients with known or suspected coronary artery disease
analysis of radiation exposure during coronary CT angiography | June 2009-
  The second specific aim is the analysis of radiation exposure during coronary CT angiography and the identification of parameters that influence radiation exposure, with the potential to provide specific guidance for interventions to lower radiation dose in the future

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Achenbach, MD, Study Chair — Universitätsklinikum Erlangen
Locations (7):
- Germany (7):
  - Kerckhoff Klinik GmbH, Bad Nauheim
  - Elisabeth Krankenhaus, Essen
  - Cardioangiologisches Centrum Bethanien, Frankfurt
  - Klinik am Eichert, Göppingen
  - Deutsches Herzzentrum München, München
  - Herzzentrum Bogenhausen, München
  - Klinikum Traunstein, Traunstein